CLINICAL TRIAL: NCT02356523
Title: Long-term Prognostic Value of Delirium in Elderly Patients With Acute Coronary Syndrome Admitted to Two Cardiac Intensive Care Units: a Prospective Study
Brief Title: Incidence and Prognostic Value of Delirium in Patients With Acute Coronary Syndromes
Status: Completed | Type: Observational
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, MD, Ospedale San Donato
Other Study IDs: Arezzo014
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delirium patients: Patients positive to Confusion Assessment Method (CAM) assessment ad admission and during hospital stay
  Interventions: Diagnostic Test: Confusion Assessment Method
- control group: Patients negative to Confusion Assessment Method (CAM) assessment ad admission and during hospital stay
  Interventions: Diagnostic Test: Confusion Assessment Method

INTERVENTIONS:
Diagnostic Test: Confusion Assessment Method — Administration of Confusion Assessment Method at patent over 65 years at admission and every day until discharge

SUMMARY:
The Purpose of this study is to evaluate the incidence of delirium in patients with acute coronary syndromes admitted to a Intensive Care Unit Patients.

DETAILED DESCRIPTION:
The present study is a prospective, two-centre registry aimed at assessing the incidence, prevalence and prognostic significance of delirium in elderly patients with acute coronary syndromes

ELIGIBILITY:
Inclusion Criteria:

* Admission in Cardiac Intensive Care Unit
* Age ≥ 65 years

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted in Cardiac Intensive Care Unit for any condition
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
diagnosis of delirium by confusion assessment method | within 24 hours of admission
  incidence of delirium in elderly patients with coronary acute syndromes

SECONDARY OUTCOMES:
adverse events incidence | 6 months
  any adverse event occurred to patients during hospital stay not due to the illness

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bolognese, MD, FESC, Study Chair — Cardiovascular Department San Donato Hospital Arezzo
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

IPD SHARING:
Plan to Share IPD: Undecided
recording in excel files

REFERENCES:
- [Background] Inouye SK. Delirium in hospitalized older patients: recognition and risk factors. J Geriatr Psychiatry Neurol. 1998 Fall;11(3):118-25; discussion 157-8. doi: 10.1177/089198879801100302. PMID 9894730
- [Background] Hsieh SJ, Ely EW, Gong MN. Can intensive care unit delirium be prevented and reduced? Lessons learned and future directions. Ann Am Thorac Soc. 2013 Dec;10(6):648-56. doi: 10.1513/AnnalsATS.201307-232FR. PMID 24364769
- [Background] McPherson JA, Wagner CE, Boehm LM, Hall JD, Johnson DC, Miller LR, Burns KM, Thompson JL, Shintani AK, Ely EW, Pandharipande PP. Delirium in the cardiovascular ICU: exploring modifiable risk factors. Crit Care Med. 2013 Feb;41(2):405-13. doi: 10.1097/CCM.0b013e31826ab49b. PMID 23263581